CLINICAL TRIAL: NCT01964378
Title: Efficacy, Safety, and Tolerability of Oral Cebranopadol Versus Morphine Sulfate PR in Subjects With Chronic Moderate to Severe Pain Related to Cancer.
Brief Title: CORAL - Cebranopadol Versus Morphine Prolonged-release in Patients With Chronic Moderate to Severe Pain Related to Cancer
Acronym: CORAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual made the study no longer feasible/decision not related to safety and efficacy
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF6005/07; 2012-001316-35 (EudraCT Number); U1111-1143-1808 (Other: World Health Organization)
Record Dates: First submitted 2013-10-07; First posted 2013-10-17 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Pain; Neoplasms; Chronic Pain
Keywords: cancer pain; neuropathic related cancer pain; morphine; cebranopadol (GRT6005); Numerical Rating Scale
MeSH Terms: conditions — Pain; Neoplasms; Chronic Pain; Cancer Pain | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cebranopadol (Experimental): Once daily oral administration. 200, 400 or 600 µg film coated tablets. Dosage 200 µg to 1000 µg per day.
  Interventions: Drug: Cebranopadol
- Morphine Prolonged Release (Active Comparator): Twice daily oral administration. 15, 30 or 45 mg morphine sulfate capsules. Dosage 30 to 150 mg per day.
  Interventions: Drug: Morphine Prolonged Release

INTERVENTIONS:
Drug: Cebranopadol — Participant will take one or two tablet(s) of cebranopadol in the morning and one or two placebo double-dummy morphine-like capsule(s) in the morning and the evening.
  Other Names: GRT6005
  Arms: Cebranopadol
Drug: Morphine Prolonged Release — Participant will take one or two morphine capsule(s) in the morning and in the evening and one or two placebo double-dummy cebranopadol-like tablet(s) in the morning.
  Arms: Morphine Prolonged Release

SUMMARY:
Pain is one of the most common symptoms associated with malignant tumor. The purpose of this trial is to determine whether cebranopadol is as effective in patients with cancer related pain as morphine sulfate prolonged release (PR).

DETAILED DESCRIPTION:
The trial comprises an enrollment period, a treatment period (titration and maintenance), and a follow-up period. Participants will receive either cebranopadol or morphine PR for 44 days. Initially participants will be titrated after 2 and then every 4 days to a morphine PR or cebranopadol dose that provides adequate analgesia and is tolerated. The titration period is planned to last 16 days. Thereafter the dose of morphine PR or cebranopadol is to be kept stable for a further 28 days, i.e. no dose adjustments will be allowed during the maintenance period. This 28 day period is the maintenance period. The follow-up period is planned for up to 18 days after the end of last pain medication treatment intake.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Negative pregnancy test before first dose.
3. Female and male participants willing to use acceptable and highly effective methods of birth control.
4. The following criteria must be fulfilled by participants:

   1. Require daily analgesia for their pain,
   2. Diagnosed with active cancer,
   3. Receiving daily opioid treatment at doses not higher than 90 mg oral morphine or its equivalent (World Health Organization Step II and Step III analgesics) for an appropriate length of time,
   4. Participants must be dissatisfied with their current pain treatment,
   5. Participants must be suffering from cancer-related but not cancer therapy-related chronic pain for a period of 4 weeks or more prior to enrollment.
5. Eastern Cooperation Oncology Group (ECOG) score 2 or below.
6. Average pain intensity over the last 24 hours of 5 or more calculated from the pain assessments recorded during the last 3 days prior to randomization.
7. Compliance with the use of the electronic diary defined as at least 3 out of 4 of the 24 hour Numerical Rating Scale entries available during the last 4 days prior to and including the day of allocation to treatment.

Exclusion Criteria:

1. Evidence of ongoing alcohol and or drug abuse and/or a history of alcohol and/or drug abuse within the last 2 years.
2. A clinically significant disease other than cancer which in the investigator's opinion may affect efficacy or safety assessments e.g., significant unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, infectious disease, psychiatric (resulting in disorientation, memory impairment or inability to report accurately) or metabolic disorders.
3. Any gastrointestinal disorder that could affect the absorption and/or elimination of Investigational Medicinal Product.
4. Any planned major surgery during the trial.
5. Known to or suspected of not being able to comply with the trial protocol and the use of Investigational Medicinal Product.
6. History of seizure disorder and/or epilepsy or any condition associated with a significant risk of seizure or epilepsy.
7. Known history and/or presence of cerebral tumor or cerebral metastases.
8. Moderate to severe hepatic impairment corresponding to Child-Pugh classification B and C. Impaired hepatic cellular integrity indicated by aspartate transaminase or alanine transaminase greater than 3 times the upper limit of normal at the Enrollment Visit.
9. Inadequate baseline bone marrow reserve with a white blood cell count below 2000/µL, a platelet count 100 000/µL or less, and a hemoglobin level below 8 g/dL at the Enrollment Visit.
10. Impaired renal function. Creatinine clearance less than 60 mL per minute(as per amendment 45 mL per minute) at the Enrollment Visit (calculated from the Cockcroft-Gault formula).
11. Forbidden concomitant medications
12. Uncontrolled hypertension
13. Clinically relevant history of hypersensitivity, allergy or contraindications to opioid medication or any of the excipients of morphine sulfate (Prolonged Released or Immediate Release), or cebranopadol film-coated tablets.
14. Chronic hepatitis B or C, or human immunodeficiency virus (HIV) known by history, or presence of active hepatitis B or C within the 3 months before the Enrollment Visit.
15. History of torsade de pointes and/or presence of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, or bradycardia).
16. Marked prolongation of corrected QT interval (Fridericia) (greater than 450 milliseconds) at the Enrollment Visit.
17. Employees of the sponsor, investigator, or trial site or family members of the employees, sponsor, or investigator.
18. Concurrent participation in another trial or planning to be enrolled in another clinical trial (i.e., administration of experimental treatment in another clinical trial) during the course of this trial.
19. Previous participation in this or other trials with cebranopadol with the following exceptions:

    * Participants who failed enrollment in this trial only because of exclusion criterion 10, and who may now be eligible can be re-enrolled.
    * Participants who failed enrollment due to technical failure of equipment (e.g., ECG machine and e-diary device).
20. Participant has received an experimental drug or used an experimental medical device within 30 days before the planned start of treatment.
21. Currently not receiving opioid treatment for cancer-related pain at the enrollment visit (i.e., opioid naïve).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Trials, Study Director — Grünenthal GmbH
Locations (42):
- AT004, Vienna, Austria
- Belgium (3):
  - BE005, Brussels
  - BE002, Ottignies
  - BE001, Sint-Niklaas
- Bulgaria (7):
  - BG001, Shumen
  - BG008, Sofia
  - BG003, Sofia
  - BG006, Sofia
  - BG007, Sofia
  - BG004, Varna
  - BG005, Vratsa
- CL005, Temuco, Chile
- HR001, Zagreb, Croatia
- Denmark (2):
  - DK006, Aalborg
  - DK004, Herlev
- Germany (2):
  - DE008, Böhlen
  - DE010, München
- Hungary (3):
  - HU004, Gyula
  - HU002, Miskolc
  - HU011, Nyíregyháza
- Poland (8):
  - PL012, Będzin
  - PL008, Bydgoszcz
  - PL013, Chorzów
  - PL014, Dąbrowa Górnicza
  - PL003, Gdansk
  - PL010, Gliwice
  - PL015, Warsaw
  - PL002, Włocławek
- Romania (4):
  - RO001, Brasov
  - RO002, Cluj-Napoca
  - RO009, Constanța
  - RO011, Craiova
- Serbia (4):
  - RS001, Belgrade
  - RS003, Belgrade
  - RS002, Kamenitz
  - RS005, Zrenjanin
- Slovakia (4):
  - SK007, Bratislava
  - SK004, Bratislava
  - SK001, Prešov
  - SK005, Pruské
- ES012, Barcelona, Spain
- UK004, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eerdekens MH, Kapanadze S, Koch ED, Kralidis G, Volkers G, Ahmedzai SH, Meissner W. Cancer-related chronic pain: Investigation of the novel analgesic drug candidate cebranopadol in a randomized, double-blind, noninferiority trial. Eur J Pain. 2019 Mar;23(3):577-588. doi: 10.1002/ejp.1331. Epub 2019 Jan 9. PMID 30365202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 29 Oct 2013 with the enrollment of the first subject and was completed on 16 Oct 2015 when the last subject completed the last follow-up examination.
Pre-assignment Details: 200 Participants were enrolled (signed consent): enrollment failures did not meet inclusion or met exclusion criteria (62 participants), died (1), withdrew consent (4), or met other reasons (1). 132 Participants were allocated to treatment and 126 were dosed (Safety Set).
Period: Overall Study
Arm/Group | Cebranopadol | Morphine Prolonged Release
Started (All allocated participants) | 66 | 66
Participants Treated (Safety Set) | 65 | 61 (4 Participants died during treatment, hereof 2 with "withdrawal..." as primary reason for discont.)
Completed | 41 | 45
Not Completed | 25 | 21
Not completed — Disc. due to death before first dosing | 0 | 1
Not completed — Disc. due to AE before first dosing | 1 | 0
Not completed — Death | 3 | 2
Not completed — Adverse Event | 12 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Inclusion/exclusion criteria not met | 1 | 3
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cebranopadol | Morphine Prolonged Release | Total
Number analyzed (Participants) | 65 | 61 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 35 | 71
  >=65 years | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.18) | 61 (10.64) | 62.4 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 38 | 39 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 58 | 60 | 118
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 65 | 61 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Romania | 2 | 1 | 3
  Hungary | 4 | 5 | 9
  Spain | 1 | 0 | 1
  Austria | 2 | 2 | 4
  Belgium | 0 | 1 | 1
  Denmark | 1 | 2 | 3
  Poland | 16 | 16 | 32
  Slovakia | 13 | 13 | 26
  Bulgaria | 7 | 4 | 11
  Chile | 2 | 0 | 2
  Serbia | 3 | 3 | 6
  Germany | 13 | 14 | 27
  Croatia | 1 | 0 | 1
Prior opioid treatment [Count of Participants; unit: Participants]
  WHO Step II analgesic | 27 | 28 | 55
  WHO Step III analgesic excluding morphine | 22 | 21 | 43
  Morphine | 16 | 12 | 28
ECOG Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status: 0 = Fully active. 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. 3 = Capable of only limited self-care. 4 = Completely disabled. 5 = Dead.
  Participants
    Status 0 | 17 | 13 | 30
    Status 1 | 30 | 30 | 60
    Status 2 | 18 | 18 | 36
    Status 3 | 0 | 0 | 0
    Status 4 | 0 | 0 | 0
    Status 5 | 0 | 0 | 0
Cancer history - Stage IV [Count of Participants; unit: Participants] — "Other" includes 10 participants (N=3 cebranopadol and N=7 morphine with an unknown stage at enrollment). Multiple entries were possible for cancer history stage thus only the details for Stage IV, the most frequent staging, is reflected.
  Participants
    Stage IV | 52 | 45 | 97
    Other | 13 | 16 | 29
Participants with a neuropathic pain component [Count of Participants; unit: Participants] — Results are based on medical history data collected.
  Participants
    Neuropathic component present | 28 | 24 | 52
    No neuropathic component present | 37 | 37 | 74
Participants with a visceral pain component [Count of Participants; unit: Participants]
  Visceral pain present | 31 | 28 | 59
  No visceral pain present | 34 | 33 | 67
Participants with a somatic pain component [Count of Participants; unit: Participants]
  Somatic pain component present | 39 | 34 | 73
  No somatic pain component present | 26 | 27 | 53
Height [Mean (Standard Deviation); unit: meter] | 1.6889 (0.09097) | 1.692 (0.07952) | 1.6904 (0.08529)
Weight [Mean (Standard Deviation); unit: kilogram(s)] | 73.52 (14.126) | 71.23 (12.807) | 72.41 (13.499)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram(s)/square meter] | 25.74 (4.39) | 24.84 (4.022) | 25.31 (4.223)
Baseline pain intensity [Mean (Standard Deviation); unit: units on a scale] — For this assessment, each participant was asked "Please rate your pain by selecting the one number that best describes your pain on average during the last 24 hours" on an 11-point Numerical Rating Scale, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The value was calculated from the mean of the 3 assessments of average pain intensity in the last 24 hours recorded during the last 3 days prior to the first dosing visit, calculated when at least one assessment in this three-day window was available.
  units on a scale | 6.23 (1.000) | 6.30 (1.230) | 6.26 (1.114)
Worst daily pain intensity [Mean (Standard Deviation); unit: units on a scale] — For this assessment, each participant was asked "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 24 hours" on an 11-point Numerical Rating Scale, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The value reported is the mean of the 3 assessments of worst pain intensity in the last 24 hours recorded during the last 3 days prior to the first dosing visit, calculated when at least one assessment in this three-day window was available.
  units on a scale | 7.27 (1.222) | 7.29 (1.117) | 7.28 (1.168)
Time since cancer pain onset [Mean (Standard Deviation); unit: weeks] — Time since cancer pain onset (in weeks) before informed consent signature.
  weeks | 62.25 (111.915) | 60.22 (79.792) | 61.27 (97.313)

OUTCOME MEASURES:

1. Primary Outcome: Average Amount of Daily Rescue Medication at the End of the Maintenance Period (Per Protocol Set)
Description: Morphine sulfate immediate release (IR) 10 mg tablets were supplied as rescue medication to trial participants. No dose adjustments of the morphine prolonged release or cebranopadol were allowed during the maintenance period. The daily use of morphine sulfate 10 mg IR tablets was documented by each participant in the trial. The total daily amount of morphine IR was subject to an upper limit recommendation. The primary endpoint is the average amount of daily rescue medication intake over the last 2 weeks of the maintenance period.
Time Frame: The last 2 weeks of the expected 6-week treatment period.
Population: The Per Protocol Set (PPS) describes a subset of subjects in the Full Analysis Set (FAS). The PPS included all allocated participants who completed at least 2 weeks of treatment in the maintenance phase and had no major protocol deviations relevant for efficacy evaluations.
Measure: Least Squares Mean (Standard Error); unit: milligram(s)/24 hours
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 43 | 45
milligram(s)/24 hours | 4.25 (1.7) | 8.92 (1.72)
Statistical Analysis 1: Comparison: Cebranopadol vs Morphine Prolonged Release; The MMRM (mixed model repeated measurement) model includes fixed effects of pooled country, treatment, week, treatment-by-week interaction, history of opioid intake, baseline pain intensity as covariate & subject-specific random effects. Dependent variable being the weekly average rescue medication intake; Test type: Non-Inferiority — Non-inferiority margin of 8 mg. Assuming equal mean values in both the cebranopadol and morphine groups, it was calculated that for the final analysis of the primary endpoint 170 subjects would have been required per treatment arm in the Per Protocol Set using a 2 sample-t-test for 90% power and a 1-sided significance level of α = 0.025; p < 0.0001, MMRM; point-estimate = -7.48, 95% CI 2-sided [-12.05 to -2.918], Standard Error of Mean 2.3

2. Primary Outcome: Average Amount of Daily Rescue Medication at the End of the Maintenance Period (Full Analysis Set)
Description: Morphine sulfate IR 10 mg tablets were supplied as rescue medication to trial participants. No dose adjustments of the morphine prolonged release or cebranopadol were allowed during the maintenance period. The daily use of morphine sulfate 10 mg IR tablets was documented by each participant in the trial. The total daily amount of morphine IR was subject to an upper limit recommendation. The primary endpoint is the average amount of daily rescue medication intake over the last 2 weeks of the maintenance period.
Time Frame: The last 2 weeks of the expected 6-week treatment period.
Population: The Full Analysis Set includes all allocated participants who took at least 1 dose of the investigational medicinal product (IMP) and had at least 1 day with information for the amount of rescue medication intake after the first intake of double-blind IMP (study drug).
Measure: Least Squares Mean (Standard Error); unit: milligram(s)/24 hours
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 64 | 61
milligram(s)/24 hours | 3.46 (1.71) | 10.94 (1.75)
Statistical Analysis 1: Comparison: Cebranopadol vs Morphine Prolonged Release; The primary endpoint will be analyzed by means of a mixed-effects model for repeated measures (MMRM), based on observed case weekly averages. Under the assumption of a missing-at-random missing data mechanism, an MMRM does not require an imputation of missing data and can obtain an improved estimate of variance; Test type: Non-Inferiority — Non-inferiority margin of 8 mg. Assuming that 65% of the participants are available for the Per Protocol Set, a total of 524 participant would have to be allocated (randomized) to IMP. With 262 participants per group in the Full Analysis Set, the non-inferiority of cebranopadol as compared to morphine sulfate prolonged release could have been demonstrated with at least 98% power and a 1-sided significance level of α = 0.025; p < 0.0001, MMRM (mixed model repeated measurement) — MMRM model: fixed effects of pooled country, treatment, week, treatment-by-week interaction, opioid intake history, baseline pain intensity as covariate & subject-specific random effects. Dependent variable: weekly average rescue medication intake; For participants with no data in the Maintenance Phase, the average amount of rescue medication over the last 3 days of titration was imputed; point-estimate = -4.67, 95% CI 2-sided [-9.245 to -0.099], Standard Error of Mean 2.3 — Non-inferiority of cebranopadol compared with morphine will be established if the upper bound of the resulting 95% confidence interval for the average treatment difference is below the non-inferiority margin of 8mg

3. Secondary Outcome: Proportion of Participants With Clinically Relevant Pain Reduction at the End of the Maintenance Period
Description: Each participant indicated the level of pain on an 11-point numerical rating scale (NRS), where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The participants entered their pain intensity in their diary on a daily basis. The pain intensity score in the 2 weeks prior to the final evaluation in the maintenance period was compared with the baseline, the baseline pain intensity was calculated based on the 3 days prior to treatment allocation.
  The definition of a clinically relevant pain reduction (yes/no) was the presence of at least 1 of the 3 following conditions:
  * Average pain intensity (i.e., average of the 24-hour pain intensities over the last 2 weeks of the Maintenance Phase) of less than 4 points on the 11-point NRS, or
  * Reduction in average pain intensity by at least 30% (compared to the baseline assessment), or
  * Reduction in average pain intensity by at least 2 points (compared to the baseline assessment).
Time Frame: The last 2 weeks of the expected 6-week treatment period.
Population: Full Analysis Set (FAS). Clinically relevant pain reduction (Yes/No) in Maintenance Week 3 and Week 4. Missing data were imputed using a multiple imputation on the weekly average pain intensity. Participants that discontinued from the trial due to a lack of efficacy were classified as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 64 | 61
Participants
  Clinically relevant pain reduction (Yes) | 48 | 51
  Clinically relevant pain reduction (No) | 16 | 10

4. Other Pre Specified Outcome: Change in Weekly Mean of the Daily Average Pain Intensity Score From Baseline
Description: Participants will be asked: "Please rate your pain by selecting the one number that best describes your pain on average during the last 24 hours." every day in the morning. They will score their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The weekly mean value of the 24-h average pain intensity will be calculated as a mean score of these daily entries of average pain intensity for each trial week.
Time Frame: Baseline; last 2 weeks of the expected 6-week treatment period
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 64 | 61
units on a scale | -3.4 (2.11) | -3.2 (1.60)

5. Other Pre Specified Outcome: Response Rate to Treatment
Description: Pain intensity will be recorded daily by each participant in the morning on an 11-point Numerical Rating Scale, ranging from 0 (no pain) to 10 (worst imaginable pain). From this, the weekly average 24-hour pain intensity will be calculated. The number of participants with a 0, 10, 20, 30, up to a 100% reduction in weekly mean pain intensity will be reported over each week and over the last 2 weeks of the maintenance period.
Time Frame: Baseline; last 2 weeks of the expected 6-week treatment period
Population: Full Analysis Set (FAS). Worsening in 24-hour pain or premature discontinuation due to lack of efficacy or Adverse Event was regarded a non-response, other missing data is imputed using last observation carried forward (LOCF).
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 64 | 61
Participants
  Non-responder | 13 | 9
  >= 0% pain reduction | 51 | 52
  >= 10% pain reduction | 50 | 52
  >= 20% pain reduction | 44 | 50
  >= 30% pain reduction | 39 | 42
  >= 40% pain reduction | 31 | 37
  >= 50% pain reduction | 26 | 27
  >= 60% pain reduction | 19 | 18
  >= 70% pain reduction | 13 | 11
  >= 80% pain reduction | 10 | 8
  >= 90% pain reduction | 5 | 2
  100% pain reduction | 3 | 2

6. Other Pre Specified Outcome: Overall Score of the Neuropathic Pain Symptom Inventory (NPSI)
Description: Participants with neuropathic pain (determined by the completion of the Douleur Neuropathique En 4 Questions [DN4] questionnaire at allocation) rated their symptoms of neuropathic pain on the Neuropathic Pain Symptom Inventory (NPSI). Ten out of 12 questions were answered on an 11-point scale 0 (no symptom present) to 10 (worst imaginable); 2 out of 12 questions assessed the duration of spontaneous pain and the number of pain attacks and were answered by selecting 1 of 5 possible responses.
  Mean scores of NPSI were calculated. The overall NPSI score was calculated by the summation of all responses in the ranges between 0 (all symptoms absent) and 1 (all symptoms present and at the worst intensity). A negative change indicates that the intensity of all the neuropathic symptom components have decreased since the start of treatment.
Time Frame: Baseline; End-of-Treatment Visit (Week 6)
Population: Subset of participants that were assessed to have Neuropathic Pain (using the DN4 questionnaire) at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 11 | 17
units on a scale | -0.15 (0.126) | -0.10 (0.129)

7. Other Pre Specified Outcome: EuroQol-5 Dimension (EQ-5D) Health Questionnaire: Weighted EQ-5D Health Status Index
Description: The EuroQol-5 Dimension Health Questionnaire is a generic health related quality of life instrument. The participants will answer 5 questions on 5 dimensions of their health related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question has 3 possible answers reflecting 3 levels of impact on the quality of life. The weighted EQ-5D health status index values are derived and reported as change from baseline. The responses to the 5 EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score (with 1 indicating "full health" and 0 representing "dead"). The higher the values (the closer the value is to 1) the better the health status in a treatment group.
  A positive change indicates an improvement.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: Full Analysis Set; means (standard deviations) are presented for the number of participants at the End-of-Treatment Visit with respective data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 49 | 52
units on a scale | 0.1 (0.331) | 0.2 (0.287)

8. Other Pre Specified Outcome: EuroQol-5 Dimension (EQ-5D) Health Questionnaire: Visual Analog Scale (VAS) Score
Description: The EuroQol-5 Dimension Health Questionnaire is a generic health related quality of life instrument. EuroQoL-5D Health State Visual Analog Scale (VAS) is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. The values indicated represent the change from the baseline, a positive value indicates an improvement.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 47 | 52
units on a scale | -0.1 (22.983) | 15.1 (24.305)

9. Other Pre Specified Outcome: Change in the Physical and Mental Component Scores From the Short Form 12® Health Survey (SF-12)
Description: The Physical and Mental Component Scores are calculated from the responses by participants to 12 questions. These 12 questions cover 8 domains, (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role participation with emotional health problems, and mental health) that a participant was asked to rate over the last week. Questions are scored on a Likert-scale.
  The Physical and Mental Component Scores were not derived as the trial was terminated.
  Changes in the individual item scores are therefore reported. A higher score indicates a better participant perceived state of health. All domains were scored on a scale from 0 (lowest level of health) to 100 (highest level of health), with 100 representing the best possible health state.
  If the values are positive there was an improvement. The higher the value the greater the improvement.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: Full Analysis Set (FAS). End of Treatment (End of Maintenance Period Visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 64 | 61
units on a scale
  Physical function: number analyzed (Participants) | 49 | 53
  Physical function | 7.1 (31.04) | 9.9 (24.68)
  Role physical: number analyzed (Participants) | 49 | 53
  Role physical | 5.1 (27.23) | 6.4 (24.10)
  Bodily pain: number analyzed (Participants) | 49 | 53
  Bodily pain | 10.2 (29.28) | 9.0 (31.43)
  General health: number analyzed (Participants) | 49 | 53
  General health | 5.4 (20.13) | 9.2 (27.38)
  Vitality: number analyzed (Participants) | 49 | 53
  Vitality | 0.0 (25.00) | 10.4 (28.77)
  Social function: number analyzed (Participants) | 49 | 53
  Social function | 7.1 (28.87) | 5.2 (33.38)
  Role emotional: number analyzed (Participants) | 49 | 53
  Role emotional | 3.3 (28.39) | 0.2 (27.57)
  Mental health: number analyzed (Participants) | 49 | 53
  Mental health | 3.1 (20.18) | 6.1 (21.32)

10. Other Pre Specified Outcome: Patient Global Impression of Change (PGIC)
Description: In the Patient Global Impression of Change (PGIC) the participant indicates the perceived change over the treatment period compared to his condition prior to the start of treatment. The participant is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: Full Analysis Set (FAS). End of Treatment (End of Maintenance Period Visit). Participants with data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 56 | 56
Participants
  Very much improved | 5 | 3
  Much improved | 18 | 17
  Minimally improved | 17 | 17
  No change | 4 | 10
  Minimally worse | 4 | 4
  Much worse | 2 | 2
  Very much worse | 0 | 0
  Missing | 6 | 3

11. Other Pre Specified Outcome: Clinical Global Impression of Change (CGIC)
Description: In the Clinical Global Impression of Change (CGIC) the clinician indicates the perceived change in patient's condition over the treatment period as compared to patient's condition prior to the start of treatment. The clinician is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: Full Analysis Set (FAS). End of Treatment (End of Maintenance Period Visit). Participants with data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 56 | 56
Participants
  Very much improved | 8 | 4
  Much improved | 20 | 26
  Minimally improved | 10 | 9
  No change | 7 | 5
  Minimally worse | 3 | 6
  Much worse | 2 | 1
  Very much worse | 0 | 2
  Missing | 6 | 3

12. Other Pre Specified Outcome: Overall Score of the Patient Assessment of Constipation Symptoms (PAC-SYM)
Description: The PAC-SYM is a 12-item self-administered questionnaire that assesses the severity of constipation-related symptoms during past 2 weeks. Items are rated on a 5-point Likert scale, where 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.The PAC-SYM contains 3 subscales: stool symptoms (5 items), abdominal symptoms (4 items), rectal symptoms (3 items). If at least 6 items are assessed, the PAC-SYM overall score is calculated as the sum of the scores of all non-missing items divided by number of non-missing items. The minimum overall score is 0, the maximum overall score is 4. If more than 6 items are missing, no overall score is calculated. Changes from baseline for the overall score are presented. If the changes in the overall (or subscale) scores are positive then there is a worsening in symptoms associated with constipation.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: Safety Set; number of participants with data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 49 | 53
units on a scale | 0.07 (0.536) | 0.07 (0.632)

13. Other Pre Specified Outcome: Change in Weekly Mean of the Daily Worst Pain Intensity Score From Baseline
Description: Participants will be asked: "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 24 hours." every day in the morning. They will score their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The weekly mean value of the 24 h worst pain intensity will be calculated as a mean score of these daily entries of worst pain intensity for each trial week. A positive change from baseline will indicate a worsening, whilst a negative change will indicate an improvement of pain.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 64 | 61
units on a scale | -3.3 (2.68) | -3.3 (2.11)

14. Other Pre Specified Outcome: Change From Baseline to End-of-Treatment Visit in Chronic Pain Sleep Inventory (CPSI) Scores
Description: The CPSI measures 5 items on 100-mm visual analog scales: trouble falling asleep (CPSI1), needing sleep medication (CPSI2), awakened by pain during the night (CPSI3) and in the morning (CPSI4) [all with anchors for 0 = never and 100 = always], and overall quality of sleep (CPSI5) [with anchors of 0 = very poor and 100 = excellent]. The sleep problem index is the sum of items CPSI1, CPSI3 and CPSI4. The minimum sleep problem index is 0 mm, the maximum 300 mm, the higher the worse. For the overall quality of sleep, minimum and maximum are 0 and 100 mm, the higher the better. A decrease in the sleep problem index indicates an improvement as does an increase in the overall quality of sleep. Changes from baseline to the End-of-Treatment Visit of the Maintenance Phase (scheduled for Week 6) were calculated.
Time Frame: Baseline; End-of-Treatment Visit (6 weeks)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol | Morphine Prolonged Release
Number analyzed (Participants) | 64 | 61
units on a scale
  Sleep Problem Index: number analyzed (Participants) | 49 | 53
  Sleep Problem Index | -62.7 (77.91) | -53.7 (77.71)
  Overall Quality of Sleep | 20.5 (36.11) | 8.1 (30.4)

ADVERSE EVENTS:
Time Frame: From first IMP intake up to day of last IMP in Week 6 + 3 weeks follow-up (max. 9 weeks in total). The All-Cause Mortality is reported for the Allocated Set. Serious and non-serious treatment emergent adverse events (i.e. events documented after the first dose of study medication and events which started before treatment and worsened after first dose of study medication) are reported for the Safety Set (all participants with at least one dose of study medication).
Arm/Group | Cebranopadol | Morphine Prolonged Release
All-Cause Mortality (participants affected / at risk) | 3/66 | 5/66
Serious Adverse Events (participants affected / at risk) | 14/65 | 11/61
Other Adverse Events (participants affected / at risk) | 52/65 | 48/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cebranopadol (N=65) | Morphine Prolonged Release (N=61)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cebranopadol (N=65) | Morphine Prolonged Release (N=61)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Somnolence (Nervous system disorders) | 6 (7) | 5 (5)
Paraesthesia (Nervous system disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 7 (7) | 10 (10)
Oedema peripheral (General disorders) | 7 (8) | 0 (0)
Asthenia (General disorders) | 6 (6) | 8 (9)
Pyrexia (General disorders) | 4 (6) | 4 (5)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (11) | 15 (15)
Nausea (Gastrointestinal disorders) | 8 (11) | 10 (12)
Vomiting (Gastrointestinal disorders) | 8 (13) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 9 (10)
Urinary tract infection (Infections and infestations) | 2 (2) | 6 (6)

LIMITATIONS AND CAVEATS:
As the enrollment was stopped for business reasons, only a fraction of the planned number of participants was enrolled; however, the trial still has a larger participant number per treatment than a majority of trials in cancer pain so far.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.